CLINICAL TRIAL: NCT01295463
Title: Descriptive Study to Evaluate the Information and Psychosocial Issues on the Risk on Infertility in Cancer Patients After Receiving Treatment in a Comprehensive Cancer Center
Brief Title: Study of Information Received About Fertility and Infertility in Patients Who Have Finished Treatment for Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Català d'Oncologia (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: ICO-FERTI; CDR0000695000 (Registry Identifier: PDQ (Physician Data Query)); EU-21105
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2011-02

CONDITIONS: Cancer
Keywords: sexual dysfunction; psychosocial effects of cancer and its treatment; infertility; colon cancer; male breast cancer; breast cancer; germ cell tumor; ovarian sarcoma; uterine sarcoma; chronic lymphocytic leukemia; osteosarcoma; chronic myelogenous leukemia; non-Hodgkin lymphoma; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); mast cell leukemia; hairy cell leukemia; prolymphocytic leukemia; adult acute lymphoblastic leukemia; adult acute myeloid leukemia; adult Hodgkin lymphoma; adult T-cell leukemia/lymphoma; small intestine lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; mycosis fungoides/Sezary syndrome; intraocular lymphoma; primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma; noncutaneous extranodal lymphoma; secondary acute myeloid leukemia; acute undifferentiated leukemia; central nervous system leukemia; T-cell large granular lymphocyte leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative; clear cell sarcoma of the kidney; Kaposi sarcoma; adult soft tissue sarcoma; chronic myelomonocytic leukemia; secondary central nervous system Hodgkin lymphoma; cutaneous lymphoma; adult non-Hodgkin lymphoma
MeSH Terms: conditions — Neoplasms; Sexual Dysfunction, Physiological; Infertility; Colonic Neoplasms; Breast Neoplasms, Male; Breast Neoplasms; Neoplasms, Germ Cell and Embryonal; Leukemia, Lymphocytic, Chronic, B-Cell; Osteosarcoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin; Congenital Abnormalities; Leukemia, Mast-Cell; Leukemia, Hairy Cell; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Hodgkin Disease; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Mycosis Fungoides; Sezary Syndrome; Intraocular Lymphoma; Leukemia, Biphenotypic, Acute; Leukemia, Large Granular Lymphocytic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Sarcoma, Kaposi; Sarcoma; Leukemia, Myelomonocytic, Chronic; Lymphoma, T-Cell, Cutaneous | interventions — Therapeutics; Psychiatric Rehabilitation

INTERVENTIONS:
Other: questionnaire administration
Other: study of socioeconomic and demographic variables
Procedure: assessment of therapy complications
Procedure: fertility assessment and management
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Learning about the amount of information on fertility and infertility by patients before they received treatment for cancer in a comprehensive cancer center may help doctors plan the best treatment.

PURPOSE: This clinical trial is studying the amount of information on fertility and infertility received by patients before treatment of cancer in patients who have finished treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the amount of information received on aspects of fertility and infertility in patients with cancer prior to receiving treatment in a comprehensive cancer center.

Secondary

* To analyze whether the information received by patients is related to the desire to be parents.
* To analyze whether the information received by patients is related to the desire to be informed.
* To determine whether there is a relationship between demographic data, diagnosis, quality of life, and associated psychosocial information received by patients.

OUTLINE: Patients complete questionnaires (Lickert and QLQ-C30) on the amount of information received prior to therapy and psychosocial issues on aspects of fertility and infertility once within 1-2 years after receiving treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer, germ cell tumor, colon cancer, leukemia, lymphoma, or sarcoma

  * Free of disease
* Completed treatment within the past 1-2 years

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Must be able to read and self-complete study questionnaires
* No psychological conditions that may prevent participation in the study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent treatment (hormonal treatment for breast cancer is allowed)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Amount of information received on aspects of fertility and infertility
Relationship between demographic data, diagnosis, quality of life, and associated psychosocial information received

CONTACTS AND LOCATIONS:
Overall Officials: Josefina Rivera, RGN, MSN, Principal Investigator — Institut Català d'Oncologia
Locations (1):
- Institut Catala D'Oncologia, L'Hospitalet de Llobregat, Spain